CLINICAL TRIAL: NCT02105883
Title: The Effect of Identification Badge on Situation Awareness During High Fidelity Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre d'apprentissage des attitudes et des habiletés cliniques (CAAHC) (Unknown)
Responsible Party: Principal Investigator, Issam Tanoubi, Université de Montréal, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MEB-2014
Record Dates: First submitted 2014-03-25; First posted 2014-04-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Patient Simulation; Awareness; Reality Testing; Residency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scenario C (control) (No Intervention): no badge
- Scenario B (badge) (Active Comparator): Use of Identification badge during scenarios (roles and places)
  Interventions: Other: Use of identification badge during scenarios

INTERVENTIONS:
Other: Use of identification badge during scenarios
  Arms: Scenario B (badge)

SUMMARY:
The purpose of this study is to evaluate if the use of identification badge (role and place) during high-fidelity simulation as an impact on situation awareness.

DETAILED DESCRIPTION:
High-fidelity simulation is well recognized as an educational tool. Mr. Issenberg completed a review(2005) that determined features of high-fidelity simulation training that lead to effective learning. It this review, it is mentioned that the validity of the simulator (realism) is essential to help learners to increase their skills and sharpen their responses. It is essential to get and maintain engagement during high-fidelity simulation and it pass by an increase in realism and situation awareness. The purpose of this study is to evaluate if the use of identification badge (physical and conceptual realism) during high-fidelity simulation as an impact on situation awareness and engagement.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiology residents (university of montreal) who participate to simulation course on crisis resources management

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Situation awareness | 2 days
  Subjects answer a 4 questions survey on situation awareness with 7 answers choices (1-strongly disagree... 7-strongly agree)
  1. I know where I was in the beginning of the scenario
  2. I know where I was during the scenario
  3. I know the role of each participant in the beginning of the scenario
  4. I Know the role of each participant during the scenario

SECONDARY OUTCOMES:
Subject's engagement in high-fidelity simulation | 2 days
  Subject answer a 2 questions survey on engagement with a 7 answers choices (1- strongly disagree...7-strongly agree)
  1. I felt emotionally concerned during the scenario
  2. The scenario was enough realistic to get engaged in the clinical situation

CONTACTS AND LOCATIONS:
Overall Officials: Issam Tanoubi, MD, Study Director — Université de Montréal; Marie-Eve Belanger, MD, Principal Investigator — Université de Montréal
Locations (1):
- CAAHC, Montreal, Quebec, Canada